CLINICAL TRIAL: NCT06450912
Title: WSI Ratio as a Biomarker for Mechanical Complication of Hemorrhagic MI
Brief Title: Novel Imaging Biomarkers for Mechanical Complications in Acute Myocardial Infarction
Acronym: MIRON-RUPTURE
Status: Completed | Type: Observational
Sponsor: Rohan Dharmakumar (Other)
Responsible Party: Sponsor-Investigator, Rohan Dharmakumar, Executive Director, Krannert Cardiovascular Research Center, Indiana University School of Medicine
Organization: Indiana University (Other)
Other Study IDs: 19978e
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Acute Myocardial Infarction; Hemorrhagic Myocardial Infarction; Myocardial Stunning; Myocardial Hemorrhage; Myocardial Reperfusion Injury; Myocardial Rupture (Post Infarct)
MeSH Terms: conditions — Myocardial Stunning; Myocardial Reperfusion Injury; Heart Rupture, Post-Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hemorrhagic Myocardial infarctions are at high risk for mechanical complications including cardiac rupture. Prediction of vulnerable myocardial segments is an important step for the stratification of hemorrhagic MI patients. Wall motion index ratio is an important parameter to determine regions of high vulnerability within the 17-segment LV model of hemorrhagic MI.

ELIGIBILITY:
Inclusion Criteria:

* Index STEMI
* Primary PCI
* Able to complete Cardiac MR - STRAIN Protocol

Exclusion Criteria:

* Contraindication to CMR (Contrast Hypersensitivity, Metallic Implants, Abnormal Rhythms, breathing difficulties)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of individuals aged 18 to 80 who have been diagnosed with acute ST-elevation myocardial infarction (STEMI) and are scheduled for emergency percutaneous coronary intervention (PCI).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Wall Strain Index for Potential Detection of Intramyocardial Hemorrhage | 48 hours Post-PCI
  Difference in Wall Strain Index values between patients with intramyocardial hemorrhage and those without, confirmed by cardiac MRI.
Wall Strain Index in Detecting the Severity of Intramyocardial Hemorrhage | 48 hours Post-PCI
  Relationship between initial Wall Strain Index measurements and the volume of intramyocardial hemorrhage quantified by cardiac MRI
Wall Strain Index Ratio in Identification of Vulnerable LV Segments for Cardiac Rupture | 48 hours Post-PCI
  Wall Strain Index Ratio for circumferential and longitudinal strain in identifying vulnerable hemorrhagic left ventricular segments at risk for rupture

CONTACTS AND LOCATIONS:
Overall Officials: Rohan Dharmakumar, PhD, Study Director — Indiana University School of Medicine; Keyur P Vora, MD FACC, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Krannert Cardiovascular Research Center, Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No